CLINICAL TRIAL: NCT03045003
Title: Testing the Feasibility and Efficacy of Two Different Intensities of an Intervention to Enhance REsilience and to Reduce SupportIve Care Needs in Cancer Patients: A Phase II TriaL
Brief Title: Testing Two Different Intensities of an Intervention to Enhance REsilience and to Reduce SupportIve Care Needs in Cancer Patients
Acronym: RESIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuela Eicher (Other)
Collaborators: ETOP IBCSG Partners Foundation (Network); Hôpital Fribourgeois (Other); University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Sponsor-Investigator, Manuela Eicher, Professeure Associée, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RESIL Trial
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Solid Tumor, Adult
Keywords: Resilience, Supportive Care, Psychosocial Care, Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Low Intensity (Other): RESIL Intervention provided by nurses and oncologists of the outpatient oncology unit.
  Interventions: Behavioral: RESIL Intervention
- Arm B: High Intensity (Other): RESIL Intervention provided by nurses and oncologists of the outpatient oncology unit plus 5 nurse-led consultations (3 face-to-face and 2 telephone consultations)
  Interventions: Behavioral: RESIL Intervention

INTERVENTIONS:
Behavioral: RESIL Intervention — Interventions tested in this study are the following: i) educational sessions with oncologists and nurses, ii) direct, electronic feed-back of resilience and needs screening in a monitoring sheet including intervention propositions and iii) consultation provided by a clinical nurse specialist to patients (in intervention B only) Interventions have been developed based on previous studies on the efficacy of screening of patient reported outcomes and direct feed-back to health care professionals and on previous studies on interventions to enhance resilience in nursing or psycho-oncology with proven efficacy. Interventions provided in the monitoring sheet have been validated by experienced Swiss oncology nurses, oncologists and psycho-oncologists.

SUMMARY:
The aim of this phase II study is to test by feasibility and efficacy of two interprofessional supportive care interventions with different intensities to facilitate resilience in patients and thereby to reduce their unmet supportive care needs.

DETAILED DESCRIPTION:
Intervention A (tested in arm A) includes screening of resilience and supportive care needs as well as direct feed-back of the screening results on a monitoring sheet to nurses and oncologists in charge of the patient. Nurses and oncologists follow three training sessions to be trained in a) resilience facilitation, b) interventions to adress supportive care needs, c) use of the monitoring sheet.

Intervention B (tested in arm B) includes same intervention as arm A supplemented by 5 structured nurse led consultations, two face to face (F2F), three by phone (PC) provided by clinical nurse specialists and based on a consultation manual.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* attending the clinic for the first chemotherapy administration
* newly diagnosed (between 4-15 weeks after diagnosis) with a new carcinoma / lymphoma
* sufficiently literate in French or German to complete questionnaires.

Exclusion Criteria:

* recurrent disease
* being treated in in-patient or palliative care units
* diagnosed with all other cancers
* in need of complex chemotherapy
* being judged by the oncologist as not being emotionally or physically capable to participate in the trial will be excluded.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Connor Davidson Resilience Scale Score Change | week 1 (first intervention application) and week 16
  Number of patients expressing a CD-RISK score change of ≥ 5 in arms A and B

SECONDARY OUTCOMES:
Supportive Care Needs Survey 9 item version score changes | week 1 (first intervention application) and week 16
  Number of patients expressing a score change in the physical and patient care needs domain and a score change of ≥ 5 in the psychological and informational needs domain of the SCNS 9 in arms A and B

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Eicher, PhD, Principal Investigator — University of Lausanne

IPD SHARING:
Plan to Share IPD: No